CLINICAL TRIAL: NCT04748003
Title: Assessment of Prevalence and Prognostic Value of Acute Myocardial Dysfunction in Severe Trauma Patients With Chest Trauma Using 2D-strain Ultrasound: A Prospective Observational Study
Brief Title: Acute Myocardial Dysfunction and Chest Trauma - The Strainy Trauma Study
Acronym: Strainy trauma
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0380
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Chest Trauma
Keywords: Severe trauma; chest trauma
MeSH Terms: conditions — Thoracic Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate whether the identification of acute myocardial dysfunction by 2D-strain transthoracic sonography in the first week following trauma would allow to better diagnose occult and severe patterns of myocardial contusion, in order to identify a subpopulation at higher risk of complications.

The measurement of myocardial strain (2D-strain) by transthoracic sonography is a robust tool to assess the myocardial function.

The investigators strongly suppose that the 2D-strain would allow to better identify subclinical MC in chest trauma, as well as the severe patterns that are associated with more organs dysfunctions and a worst outcome.

DETAILED DESCRIPTION:
Thoracic trauma is the cause of significant morbidity and accounts for 25% of trauma-related deaths.

The myocardial contusion (MC) is a distinct injury, which has a prevalence increasing with the severity of the trauma. The diagnostic tool is a major factor to vary the prevalence of MC (i.e. clinical exam, biology, electrocardiogram), with the highest values for autopsy series, until 24% of patients. It does not exist therefore of gold standard for the diagnosis of MC in clinical practice leading to a modest knowledge of this nosological entity. In clinical practice, troponin plasma level determines the diagnostic.

Otherwise, the measurement of myocardial strain (2D-strain) by transthoracic echocardiography (TTE) is a robust tool to assess the myocardial function. This ultrasound analysis allows an objective and topographical quantification of an acute myocardial dysfunction, be it global or segmental. 2D-strain has been thus has been validated for the diagnosis of myocardial dysfunction in medical setting. Its use in trauma setting has never been reported.

ELIGIBILITY:
Inclusion Criteria:

* severe trauma patients with blunt chest trauma
* (AIS Thorax score ≥ 1)
* admitted in our trauma intensive care unit
* and included within the 24 first hours following trauma

Exclusion Criteria:

* Imminent death
* Recovered cardiocirculatory arrest following trauma
* Critical patient : AIS score ≥5 on 1 lesion, requiring ECLS (extracorporeal life support) or REBOA (resuscitative endovascular balloon occlusion of the aorta)
* Refractory hypovolaemia
* Arrhythmia, atrial fibrillation
* Congenital heart disease, ischemic cardiomyopathy, moderate or severe pre-existing valvular heart disease, pulmonary arterial hypertension (PAH)
* Valve prosthesis or pacemaker
* Insufficient quality of ultrasound image to allow correct assessment of 2D-strain
* Pregnant woman and underage patients

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe trauma patients with blunt chest trauma
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-02-28 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Occurrence of an a segmental or global acute myocardial dysfunction | In the first week following trauma
  Using transthoracic echocardiography to assess the myocardial function

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan CHARBIT, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, Montepllier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC